CLINICAL TRIAL: NCT00714662
Title: Effects of Different Frequencies of High-Flux Membranes on Blood Pressure, Fluid Balance, and Indices of Nutrition, Inflammation, and Dialysis Adequacy in Chronic Hemodialysis Patients - Comparisons Between Thrice vs Once Weekly
Brief Title: High Flux Hemodialysis Thrice Versus Once
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Mrs. Hsiu-Chin Lee Kidney Research Fund (Unknown)
Responsible Party: Yung-Ming Chen/M.D., National Taiwan University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200803055R
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: End-Stage Renal Disease
Keywords: high flux hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: high flux hemodialyzer (FX-60, FX-80 or FX-100) — three sessions per week
  Other Names: FX-60, FX-80 or FX-100

SUMMARY:
To investigate the influence of different dialysis frequencies on the outcome of end-stage renal disease patients undergoing chronic hemodialysis therapy.

DETAILED DESCRIPTION:
This study will be conducted in the HD center at NTUH. Patients undergoing chronic HD for at least 6 months will be evaluated for eligibility. Patients with previous adverse reactions to FX series dialyzer will not be included in this study. Detailed demographic physical characteristics of the participants will be recorded, including age, gender, underlying diseases, blood pressure, intradialytic complications, as well as indices of nutrition, inflammation, and dialysis adequacy. Eligible patients will first undergo a 4-week run-in HD with conventional-flux dialyzer twice weekly plus high-flux dialyzer once weekly (i.e., basic formula), followed by random allocation into two separate groups. Patients in group A will continue HD with the basic formula, while those in group B will receive HD using high-flux membranes thrice weekly. Three months later, all participants will be put back on HD with basic formula for 1 month (wash-out period). Group A patients will then be switched to receive HD with high-flux membranes thrice weekly, and group B patients will be changed to undergo HD with basic formula for another 3 months. Laboratory tests will include monthly biochemistry and hemogram, plus blood and urine specimens taken on 4 occasions before and during the study (baseline, end of the first 3 months, end of wash-out, and end of the second 3 months) to investigate selective markers and indices for nutrition, inflammation, and dialysis adequacy.

ELIGIBILITY:
Inclusion Criteria:

1. ESRD patients under regular thrice weekly HD for more than 3 months in NTUH HD center.
2. Age: 18~80 years old.
3. Blood flow during dialysis ≧ 250ml/min

Exclusion Criteria:

1. Previous allergy to heparin or FX series dialyzer (FX-60, FX-80, FX-100)
2. Pre-dialysis systolic blood pressure ≦ 100mmHg (2week prior to enrollment)
3. Bacteremia, myocardial infarction or stroke in previous 3 months.
4. Known diagnosis with dialysis related amyloidosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-02 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
blood pressure, fluid balance, and indices of nutrition, inflammation, and dialysis adequacy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Ming Chen, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan